CLINICAL TRIAL: NCT00787969
Title: Phase I/II Trial of Rituximab, Cladribine, and Temsirolimus (RCT) Therapy in Newly Diagnosed Mantle Cell Lymphoma (MCL)
Brief Title: Rituximab, Cladribine, and Temsirolimus in Treating Patients With Newly Diagnosed Mantle Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N078D; NCI-2009-00669 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000619329 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Lymphoma
Keywords: stage I mantle cell lymphoma; Stage II Contiguous Mantle Cell Lymphoma; Stage II Non-Contiguous Mantle Cell Lymphoma; Stage III Mantle Cell Lymphoma; Stage IV Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Rituximab; Cladribine; temsirolimus; Filgrastim; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (rituximab, cladribine, temsirolimus) (Experimental): Patients receive rituximab IV on day 1 and cladribine IV over 2 hours on days 1-5. Patients then receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Patients also receive filgrastim SC on days 6-15 or pegfilgrastim SC on day 6. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Drug: cladribine; Drug: temsirolimus; Biological: Filgrastim; Biological: Pegfilgrastim

INTERVENTIONS:
Biological: rituximab — Give IV
Drug: cladribine — Give IV
Drug: temsirolimus — Give IV
Biological: Filgrastim — Give SC
Biological: Pegfilgrastim

SUMMARY:
This phase I/II trial studies the side effects and best dose of temsirolimus when given together with cladribine and rituximab and to see how well it works in treating patients with newly diagnosed mantle cell lymphoma. Monoclonal antibodies, such as rituximab, may interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as cladribine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Temsirolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving temsirolimus together with cladribine and rituximab may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy and safety of the combination of rituximab, cladribine, and temsirolimus for newly diagnosed mantle cell lymphoma.

II. To determine the maximum tolerated dose (MTD) of temsirolimus combined with a fixed dose and schedule of rituximab and cladribine. (Phase I) III. To assess the efficacy of the combination of rituximab, cladribine, and temsirolimus for newly diagnosed mantle cell lymphoma with the proportion of complete responses as the primary endpoint. (Phase II)

SECONDARY OBJECTIVES:

I. To assess other measures of efficacy of the regimen including progression free survival, duration of response, and overall survival.

II. To assess the toxicity profile of the combination of rituximab, cladribine, and temsirolimus.

III. To assess efficacy using traditional lymphoma parameters and absolute lymphocyte count.

IV. To assess metabolic markers (hyperglycemia, hyperlipidemia) as markers of mammalian target of rapamycin (mTOR) inhibition using the glucose and lipid measurements being performed in the clinical laboratory as part of routine care.

V. To correlate response with serum free light chains, single nucleotide polymorphisms (SNPs) in host immune genes, vitamin D metabolites, and phosphatidylinositide 3-kinase (PI3K) pathway member expression.

VI. As part of ongoing research for North Central Cancer Treatment Group (NCCTG) lymphoma studies, paraffin-embedded tissue blocks/slides and blood products will be banked for future studies.

OUTLINE: This is a phase I, dose-escalation study of temsirolimus followed by a phase II study.

Patients receive rituximab intravenously (IV) on day 1 and cladribine IV over 2 hours on days 1-5. Patients then receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Patients also receive filgrastim subcutaneously (SC) on days 6-15 or pegfilgrastim SC on day 6. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 4 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed mantle cell lymphoma (MCL); the diagnosis must be confirmed by NCCTG pre-registration pathology review by Dr. Paul Kurtin or his designate; it is recommended that the biopsy be an excisional biopsy, but adequate core-needle biopsies will be accepted as long as they are considered adequate for registration by Dr. Kurtin or his designate; the tumor must be cyclin D-1 positive by immunohistochemistry or have evidence of a t(11;14) translocation by fluorescence based in situ hybridization (FISH) or cytogenetics
* Measurable or assessable disease, defined as at least one of the following:

  * A lymph node or tumor mass that is >= 2.0 cm in at least one dimension by positron emission tomography (PET)/computed tomography (CT), CT, magnetic resonance imaging (MRI), or plain radiograph imaging
  * Splenic enlargement may be used as a measurable parameter if the spleen is palpable >= 3 cm below the left costal margin
  * Diffuse infiltration of an organ such as the stomach, bone marrow, peripheral blood, liver, lungs, or bowel by lymphoma without a discrete mass would constitute assessable, but not measurable, disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, 2, or 3
* Life expectancy >= 12 weeks
* Absolute neutrophil count (ANC) >= 1,500/mm³
* Platelet count (PLT) >= 100,000/mm³
* Serum creatinine =< 2.0 mg/dL
* Serum total bilirubin (or direct bilirubin if total is abnormal) =< institutional upper limit of normal (ULN) with or without secondary liver involvement
* Serum glutamic oxaloacetic transaminase (SGOT) =< 3 x institutional ULN (exception: if there is liver involvement, SGOT must be =< 5 x institutional ULN)
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Willingness to return to NCCTG enrolling institution for follow-up
* Willingness to provide the blood specimens as required by the protocol
* Willingness to provide tissue specimens as required by the protocol
* Willing to return to NCCTG enrolling institution for follow-up
* Willing to provide blood and tissue specimens as required by the protocol
* Willing to abstain from eating grapefruit or drinking grapefruit juice
* Willingness to abstain from eating grapefruit or drinking grapefruit juice for the duration of the study

Exclusion Criteria

* Any prior therapy for mantle cell non-Hodgkin lymphoma including radiation therapy; exception: patient may have undergone a splenectomy for diagnosis, cytopenia, or systematic splenomegaly
* Active or uncontrolled infection
* Any of the following cardiac conditions:

  * Uncontrolled high blood pressure
  * Unstable angina
  * Active congestive heart failure
  * Myocardial infarction =< 6 months
  * Serious uncontrolled cardiac arrhythmia
* Known central nervous system (CNS) involvement
* Any of the following:

  * Pregnant women or women of reproductive ability who are unwilling to use effective contraception while taking the drug and for 12 months after stopping treatment
  * Nursing women
  * Men who are unwilling to use a condom (even if they have undergone a prior vasectomy) while having intercourse with any woman, while taking the drug and for 12 months after stopping treatment
* Medical or psychiatric conditions which, in the opinion of the investigator, make the patient a poor risk for participation
* Known to be human immunodeficiency virus (HIV) positive; HIV testing is not required but should be done if clinically indicated; HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study
* Concurrent malignancy =< 5 years ago; exceptions: carcinoma in situ of the cervix, resected basal cell or squamous cell carcinomas of the skin, or prostate cancer that is in remission following a radical retropubic prostatectomy or radiation therapy; if there is a history of prior malignancy, they must not be receiving other specific treatment (other than hormonal therapy) for their cancer
* Known hypersensitivity to rituximab or its components, or to murine proteins
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Prior treatment with an mTOR inhibitor
* Autologous or allogeneic stem cell transplant planned as part of initial therapy
* Receiving enzyme-inducing antiepileptic drugs (enzyme inducing anti-epileptic drugs [EIAEDs]; e.g., phenytoin, fosphenytoin, carbamazepine, oxcarbazepine, phenobarbital, or primidone); any other potent cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inducer such as rifampin, glucocorticoids at greater than adrenal replacement levels, or St. John's wort; or receiving strong CYP3A4 inhibitors * Note: if these agents are discontinued, temsirolimus therapy can begin >= 7 days after discontinuation of such agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2009-04 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Number of dose limiting toxicity incidents as per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 3.0 (Phase I) | 28 days
Proportion of complete tumor responses defined as complete remission (CR) as the objective status (Phase II) | Up to 5 years

SECONDARY OUTCOMES:
Overall survival | up to 5 years
Progression-free survival (PFS) | up to 5 years
Time to disease progression | up to 5 years
Duration of response, defined as date at which the patient's objective status is first noted to be either a CR or partial remission to the date progression is documented | Up to 5 years
Survival time | Up to 5 years
Frequency and severity of adverse events assessed by CTCAE v3.0 | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: David J. Inwards, MD, Study Chair — Mayo Clinic
Locations (144):
- United States (144):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - Michiana Hematology Oncology PC - Niles, Niles, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Derived] Inwards DJ, Fishkin PA, LaPlant BR, Drake MT, Kurtin PJ, Nikcevich DA, Wender DB, Lair BS, Witzig TE. Phase I trial of rituximab, cladribine, and temsirolimus (RCT) for initial therapy of mantle cell lymphoma. Ann Oncol. 2014 Oct;25(10):2020-2024. doi: 10.1093/annonc/mdu273. Epub 2014 Jul 23. PMID 25057177